CLINICAL TRIAL: NCT04054986
Title: Phase 1 Study Using First-in-Human Acidosis Imaging With [18F]AlF-cysVar3 pHLIP® (18F-Var3) in Patients With Breast Cancer for Determination of Safety, Biodistribution and Radiation Dosimetry
Brief Title: Study of the Imaging Agent 18F-Var3 in Patients With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-147
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; 18F-Var3; First in human; Acidosis imaging; Memorial Sloan Kettering Cancer Center; 19-147
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Breast Cancer (Experimental): Breast cancer
  Interventions: Diagnostic Test: F-Var3 PET/CT; Other: Blood draw

INTERVENTIONS:
Diagnostic Test: F-Var3 PET/CT — Participants will undergo up to 5 serial F-Var3 PET/CT scans within 25 minutes of the injection of 18F-Var3, 30, 60, 120 and 240 minutes after injection of the 18FVar3.
Other: Blood draw — Collection of blood for research tests before the injection, 30, 60, 120 and 240 min after the injection.

SUMMARY:
The purpose of this study is to measure the safety of the investigational imaging agent, 18F-Var3 and to determine if it is helpful in providing information about how tumor tissues behave.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Biopsy-proven breast malignancy
* >/= 1 viable lesion, >/= 1 cm, confirmed on CT, MR, or FDG PET/CT within 4 weeks of protocol enrollment
* Newly diagnosed or recurrent disease, on or off therapy
* ECOG performance of 0-2 *Note: Lesions are considered viable if they are stable or increasing soft tissue lesions, or if they are FDG-avid bone lesions

Exclusion Criteria:

* Life expectancy < 3 months
* Pregnancy or lactation
* Biopsy or other surgical procedures within 48 hours prior to receiving study intervention
* Patients who cannot undergo PT/CT scanning because of weight limits. PET/CT scanners may not be able to function with patients over 400 pounds

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5.0 | 30 days after completion of study treatment and assessments
  The safety of patients will be evaluated using Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Grade 1 and grade 2 toxicities are considered safe.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Riedle, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org